CLINICAL TRIAL: NCT05986799
Title: A Randomized, Controlled Trial of Efficacy of Amway Herbal Drink to Improve Skin Anti-aging
Brief Title: The Efficacy of Amway Herbal Drink to Improve Skin Anti-aging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amway (China) R&D Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 23-RD-05-AY-001
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Skin Laxity; Skin Lines
Keywords: Anti-aging; Amway herbal drink
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amway Herbal Drink (Active Comparator): Amway Herbal Drink: 5g/sachet, containing the following active ingredients:
  * Extract of Phyllanthus emblica
  * Sophora flower extract
  * Wild cherry extract
  * Flower extract of Dendrobium candidum
  * Pomegranate extract
  * Resistant dextrin
  * γ-cyclodextrin
  Interventions: Dietary Supplement: Amway Herbal Drink
- Placebo Drink (Placebo Comparator): Placebo Drink: 5g/sachet, containing the following active ingredients:
  * Maltodextrin
  * Sugar
  * Honey
  Interventions: Dietary Supplement: Placebo Drink

INTERVENTIONS:
Dietary Supplement: Amway Herbal Drink — 1 sachet per time, 3 times daily, for 3 months period.
  Arms: Amway Herbal Drink
Dietary Supplement: Placebo Drink — 1 sachet per time, 3 times daily, for 3 months period.
  Arms: Placebo Drink

SUMMARY:
This goal of this two arms, randomized, double-blind controlled trial is to study whether Amway herbal drink could improve skin anti-aging in the middle-aged people of 30-60 years old. The main questions it aims to answer are:

1. whether skin elasticity will be improved measured by Cutometer
2. whether skin wrinkles/roughness/pores will be improved measured by Antera 3D

30 eligible Participants will be enrolled in one center and randomly assigned to two study groups (Amway herbal drink group and placebo drink group). Up to four study visits will be made by the subject over a 3-month period intervention and all clinical data will be captured and recorded into CTMS (Clinical Trial Management System) for data analysis and reporting.

Researchers will compare Amway herbal drink group and placebo drink group to see if consumption of Amway herbal drink could significantly improve skin anti-aging at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, aged 30 to 60 years, with a gender ratio of 3:7;
* Subjects are healthy;
* Visual assessment, smoothness is greater than or equal to 3 points (according to the Test Method of Efficacy Measurement of Nourishing Cosmetic Products issued by Chinese Association of Fragrance Flavor and Cosmetic Industries, the smaller the index, the better. Please refer to appendix II);
* Visual assessment, the gloss index is greater than or equal to 4 points (according to the Unilever Radiance Scale, the smaller the index is the better. Please refer to appendix III);
* Subjects could not use facial whitening and moisturizing products during the trial;
* Agree not to take other oral products with similar efficacy (such as collagen, sodium hyaluronate, etc.) during the trial. During the trial, participants agreed not to take any drugs or supplements. Do not do any medical beauty projects during the trial, do not participate in other interventional clinical research;
* Have a full understanding of the purpose, benefits, and possible risks and side effects of the study;
* Willing to comply with all research requirements and procedures;
* Understand the test procedure, read, and sign an appropriate Informed Consent Form indicating their willingness to participate.

Exclusion Criteria:

* Use of any medications or supplements that may alter skin properties during the first 3 months of enrollment;
* Skin disease patients;
* Ggastrointestinal symptoms being treated;
* Lactose intolerance, allergy to fish and its products;
* Present with other organic diseases that affect intestinal function, such as history of gastrointestinal resection, colon or rectal cancer, inflammatory bowel disease, diabetes, hyperthyroidism or hypothyroidism, congenital megacolon, scleroderma, anorexia nervosa, etc.;
* Controlling diet, exercising more, or taking medications to control weight or affect appetite in the last 3 months;
* Subjects have any of the following medical history or clinical findings that may affect the evaluation of the trial effect: significant gastrointestinal disorders, liver, kidney, endocrine, hematological, respiratory and cardiovascular diseases;
* Abuse of alcohol or other illicit drugs, supplements currently or in the past, or OTC prescription drugs that may cause intestinal dysfunction or interfere with the evaluation of trial effects;
* Frequent use of drugs that may affect gastrointestinal function or the immune system, as judged by the researcher;
* Use of laxatives or other digestive substances in the 2 weeks prior to trial commencement;
* Women who are pregnant or breastfeeding, or who plan to become pregnant during the trial;
* PI considers that volunteers cannot fully cooperate with the trial arrangement.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-13 (Estimated); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Change of Skin Elasticity | baseline day 0, day 90
  The changes of skin elasticity from baseline to day 90 by CK Cutometer MPA580

SECONDARY OUTCOMES:
Change of Facial Lines/Wrinkles | baseline day 0, day 45, day 90
  The changes of facial lines/wrinkles by Miravex Antera 3D imaging system

CONTACTS AND LOCATIONS:
Overall Officials: Yun Wang, MD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ai You Mei Medical Beauty Clinic, Jinhua, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cao C, Xiao Z, Wu Y, Ge C. Diet and Skin Aging-From the Perspective of Food Nutrition. Nutrients. 2020 Mar 24;12(3):870. doi: 10.3390/nu12030870. PMID 32213934
- [Background] Blanpain C, Fuchs E. Epidermal stem cells of the skin. Annu Rev Cell Dev Biol. 2006;22:339-73. doi: 10.1146/annurev.cellbio.22.010305.104357. PMID 16824012
- [Background] Zhang S, Duan E. Fighting against Skin Aging: The Way from Bench to Bedside. Cell Transplant. 2018 May;27(5):729-738. doi: 10.1177/0963689717725755. Epub 2018 Apr 25. PMID 29692196
- [Background] Blume-Peytavi U, Kottner J, Sterry W, Hodin MW, Griffiths TW, Watson RE, Hay RJ, Griffiths CE. Age-Associated Skin Conditions and Diseases: Current Perspectives and Future Options. Gerontologist. 2016 Apr;56 Suppl 2:S230-42. doi: 10.1093/geront/gnw003. PMID 26994263
- [Background] Michalak M. Plant-Derived Antioxidants: Significance in Skin Health and the Ageing Process. Int J Mol Sci. 2022 Jan 6;23(2):585. doi: 10.3390/ijms23020585. PMID 35054770
- [Background] Fam VW, Charoenwoodhipong P, Sivamani RK, Holt RR, Keen CL, Hackman RM. Plant-Based Foods for Skin Health: A Narrative Review. J Acad Nutr Diet. 2022 Mar;122(3):614-629. doi: 10.1016/j.jand.2021.10.024. Epub 2021 Oct 30. PMID 34728412
- [Background] Chaikul P, Kanlayavattanakul M, Somkumnerd J, Lourith N. Phyllanthus emblica L. (amla) branch: A safe and effective ingredient against skin aging. J Tradit Complement Med. 2021 Feb 9;11(5):390-399. doi: 10.1016/j.jtcme.2021.02.004. eCollection 2021 Sep. PMID 34522633
- [Background] Binic I, Lazarevic V, Ljubenovic M, Mojsa J, Sokolovic D. Skin ageing: natural weapons and strategies. Evid Based Complement Alternat Med. 2013;2013:827248. doi: 10.1155/2013/827248. Epub 2013 Jan 29. PMID 23431351
- [Background] Lee HR, Ryu HG, Lee Y, Park JA, Kim S, Lee CE, Jung S, Lee KH. Effect of Aronia Extract on Collagen Synthesis in Human Skin Cell and Dermal Equivalent. Oxid Med Cell Longev. 2022 Aug 8;2022:4392256. doi: 10.1155/2022/4392256. eCollection 2022. PMID 35979399
- [Background] Benatrehina PA, Pan L, Naman CB, Li J, Kinghorn AD. Usage, biological activity, and safety of selected botanical dietary supplements consumed in the United States. J Tradit Complement Med. 2018 Mar 2;8(2):267-277. doi: 10.1016/j.jtcme.2018.01.006. eCollection 2018 Apr. PMID 29736381
- [Background] Zhou H, Zhou L, Li B, Yue R. Anti-cyclooxygenase, anti-glycation, and anti-skin aging effect of Dendrobium officinale flowers' aqueous extract and its phytochemical validation in aging. Front Immunol. 2023 Mar 17;14:1095848. doi: 10.3389/fimmu.2023.1095848. eCollection 2023. PMID 37006297